CLINICAL TRIAL: NCT07332533
Title: A Phase II/III Study of KN026 Combined Chemotherapy With or Without Enlonstobart as First-line Treatment in HER2-positive Unresectable Locally Advanced or Metastatic Gastric Cancer.
Brief Title: A Study of KN026-based Combination Therapy in HER2-positive Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN026-006
Record Dates: First submitted 2025-12-25; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Trastuzumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, controlled, multi-center Phase II/III clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A：Combination of KN026 and CAPOX/PF with or without enlonstobart (Experimental)
  Interventions: Drug: KN026; Drug: Capecitabine; Drug: Enlonstobart; Drug: Oxaliplatin; Drug: Cisplatin; Drug: Fluorouracil
- Group B: Combination of trastuzumab, and CAPOX/PF with or without enlonstobart (Experimental)
  Interventions: Drug: Capecitabine; Drug: Enlonstobart; Drug: Oxaliplatin; Drug: Trastuzumab; Drug: Cisplatin; Drug: Fluorouracil
- Experimental group: Combination of KN026 and CAPOX/PF with or without enlonstobart (Experimental)
  Interventions: Drug: KN026; Drug: Capecitabine; Drug: Enlonstobart; Drug: Oxaliplatin; Drug: Cisplatin; Drug: Fluorouracil
- Control group：Combination of trastuzumab and CAPOX/PF with or without Pembrolizumab (Experimental)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Trastuzumab; Drug: Pembolizumab; Drug: Cisplatin; Drug: Fluorouracil

INTERVENTIONS:
Drug: KN026 — In accordance with the protocol
  Arms: Experimental group: Combination of KN026 and CAPOX/PF with or without enlonstobart; Group A：Combination of KN026 and CAPOX/PF with or without enlonstobart
Drug: Capecitabine — Capecitabine is for oral administration.
Drug: Enlonstobart — Enlonstobart is administered by intravenous infusion.
  Arms: Experimental group: Combination of KN026 and CAPOX/PF with or without enlonstobart; Group A：Combination of KN026 and CAPOX/PF with or without enlonstobart; Group B: Combination of trastuzumab, and CAPOX/PF with or without enlonstobart
Drug: Oxaliplatin — Oxaliplatin is administered by intravenous infusion.
Drug: Trastuzumab — Trastuzumab is administered by intravenous infusion.
  Arms: Control group：Combination of trastuzumab and CAPOX/PF with or without Pembrolizumab; Group B: Combination of trastuzumab, and CAPOX/PF with or without enlonstobart
Drug: Pembolizumab — Pembolizumab is administered by intravenous infusion.
  Arms: Control group：Combination of trastuzumab and CAPOX/PF with or without Pembrolizumab
Drug: Cisplatin — Cisplatin is administered by intravenous infusion.
Drug: Fluorouracil — Fluorouracil is administered by intravenous infusion.

SUMMARY:
This study is designed to compare the efficacy and safety of KN026 combined chemotherapy with or without Enlonstobart versus Trastuzumab combined chemotherapy with or without Pembrolizumab as first-line treatment in HER2-positive unresectable locally advanced or metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Age≥18 years old.

* Histologically or cytologically confirmed diagnosis of gastric cancer.
* Participants unresectable locally advanced or metastatic gastric cancer who had not received systemic treatment (participants who had progressed 6 months after prior neoadjuvant/adjuvant therapy could be enrolled).
* Confirmed to be HER2 positive (HER2-positive is defined as IHC 3+ or IHC 2+ with ISH positive) and PD-L1 status (participants of phase III should be confirmed by the pathology department of participating study center).
* Phase II: Presence of at least 1 measurable lesion per RECIST 1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Phase III:Presence of at least 1 evaluable lesion per RECIST 1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* ECOG PS of 0 - 1.
* Expected survival ≥ 3 months.
* Participants with adequate organ functions.
* Female and male participants of childbearing age agree to take adequate contraceptive measures during and upon completion of the study for 7 months after the last dose. Female participants of childbearing age must have a negative blood pregnancy test within 7 days before randomization.
* Voluntarily agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Has received anti-tumor treatment such as systemic chemotherapy or other trial interventions within 28 days, or immunotherapy (e.g. interleukin, interferon, thymospipeptide, etc.), hormone therapy or targeted therapy within 14 days or 5 half-life (whichever is shorter) before randomization.
* Participants with brain metastasis or spinal cord compression at screening (except for completed local treatment and discontinued glucocorticoids for at least 4 weeks before randomization , and stable central nervous system imaging and brain metastasis symptoms for at least 4 weeks).
* Participants with PD-L1 CPS ≥1, who are receiving long-term immunotherapy (e.g., cyclosporine) or require daily systemic steroid therapy (e.g., >20 mg prednisone or equivalent), except those who treated with local glucocorticoids using nasal spray, inhalation, or other pathways.
* Participants with PD-L1CPS ≥1, who have an active autoimmune disease or have a history of autoimmune disease 2 years before randomization and still require systemic treatment. However, participant with the following diseases is allowed to enroll: well-controlled type I diabetes, well-controlled hypothyroidism that requires hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss), or participant who is expected to not recur without external triggers.
* Participate in another clinical trial, unless it is an observational (non-intervention) clinical trial or is in the follow-up period of an intervention trial.
* Participants who have undergone major surgery or had invasive intervention within 28 days before randomization. Or those who plan to undergo systematic or local tumor resection during the trial .
* Any Chinese patent medicine with anti-cancer activity approved by the National Drug Administration (regardless of cancer type) has been used within 14 days before randomization.
* Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
* Active bacterial, fungal or viral infection before randomization. Participant who has recieved preventive infection treatment but has no clinical manifestations before randomization could be considered to enroll.
* Has a history of immunodeficiency, including HIV-positive.
* Active hepatitis B or C infection. Participant with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) need to test Hepatitis B virus DeoxyriboNucleic Acid (HBV-DNA), and HBV-DNA is higher than 500 IU/mL (or 2500 copies/ml) ; Participants with positive for hepatitis C (HCV) antibody and whose Hepatitis C virus Ribonucleic Acid (HCV-RNA) is higher than 1000 copies/ml or UNL (whichever is lower).
* Has a history of tuberculosis treatment within 2 years before randomization.
* Has activity or a history of interstitial lung disease at any stage and/or pulmonary function injury, a history of interstitial pneumonia requiring hormone therapy, or the imaging cannot rule out suspected interstitial lung disease/pneumonia at screening.
* Known to have low activity or lack of dihydropyrimidine dehydrogenase (DPD).
* Participants with peripheral neuropathy of grade > 1.
* Participants with clinically significant gastrointestinal diseases including but not limited to severe liver diseases, ulcerative colitis, Crohn's disease and other gastrointestinal diseases 28 days before randomization; Unable to swallow orally, or there are conditions that have been judged by researchers to seriously affect gastrointestinal absorption (such as malabsorption syndrome, etc.).
* Has a history of severe cardiovascular disease.
* History of any other malignant tumors within 5 years before randomization.
* pleural effussion, peritoneal dropsy or pericardial effusion requiring drainage within 2 weeks before randomization.
* Live vaccination within 28 days before randomization. Note: Seasonal influenza vaccine is a broadly inactivated vaccine and is allowed to be used;
* Breastfeeding women.
* Otherwise considered inappropriate for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 490 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by investigator in Phase II | Up to approximately 5 years
Progression-Free Survival (PFS) by BIRC in Phase III | Up to approximately 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) in Phase III | Up to approximately 5 years